CLINICAL TRIAL: NCT05840172
Title: An Open Label, Randomised, 3-way Cross-over, Single-centre, Clinical Investigation to Evaluate the Effectiveness of Benzocaine in Two NRL Condoms Compared With a Standard NRL Control Without Benzocaine in Prolonging Time to Ejaculation in Healthy Adult Men Who Feel They Ejaculate Too Quickly During Vaginal Sex
Brief Title: A Clinical Investigation to Assess the Effectiveness of Benzocaine in NRL Condoms in Healthy Adult Men Who Feel They Ejaculate Too Quickly During Vaginal Sex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 5078401
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Ejaculation Delayed
MeSH Terms: conditions — Ejaculatory Dysfunction

STUDY DESIGN:
Intervention Model Description: The condom types will be tested in a 3-way cross-over design where subjects will be randomised to use each of the 3 condom types in a defined order, according to the randomisation schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test condom A (NRL condom with 5% benzocaine paste) (Experimental): Following randomization, each subject will be given one set of 8 condoms as per randomisation schedule. After reporting at least 4 duration records (from vaginal entry to ejaculation), subjects will return to the clinical site for collection of their next set of condoms.
  Interventions: Device: Test condom A (NRL condom with 5% benzocaine paste)
- Test condom B (NRL condom with 3% benzocaine paste) (Experimental): Following randomization, each subject will be given one set of 8 condoms as per randomisation schedule. After reporting at least 4 duration records (from vaginal entry to ejaculation), subjects will return to the clinical site for collection of their next set of condoms.
  Interventions: Device: Test condom B (NRL condom with 3% benzocaine paste)
- Control NRL condom (Placebo Comparator): Following randomization, each subject will be given one set of 8 condoms as per randomisation schedule. After reporting at least 4 duration records (from vaginal entry to ejaculation), subjects will return to the clinical site for collection of their next set of condoms.
  Interventions: Device: Control NRL condom

INTERVENTIONS:
Device: Test condom A (NRL condom with 5% benzocaine paste) — In each assessment period, subjects will be provided with a condom type to use during vaginal intercourse and will report at least 4 duration records (from vaginal entry to ejaculation) over a 4-week period. Subjects will repeat the assessment period each to test all 3 condom types.
  Arms: Test condom A (NRL condom with 5% benzocaine paste)
Device: Test condom B (NRL condom with 3% benzocaine paste) — In each assessment period, subjects will be provided with a condom type to use during vaginal intercourse and will report at least 4 duration records (from vaginal entry to ejaculation) over a 4-week period. Subjects will repeat the assessment period each to test all 3 condom types.
  Arms: Test condom B (NRL condom with 3% benzocaine paste)
Device: Control NRL condom — IIn each assessment period, subjects will be provided with a condom type to use during vaginal intercourse and will report at least 4 duration records (from vaginal entry to ejaculation) over a 4-week period. Subjects will repeat the assessment period each to test all 3 condom types.
  Arms: Control NRL condom

SUMMARY:
The investigation is to evaluate the effectiveness of benzocaine in two NRL condoms compared with a standard NRL control without benzocaine in prolonging time to ejaculation in healthy adult men who feel they ejaculate too quickly during vaginal sex.

DETAILED DESCRIPTION:
In this investigation, two NRL condoms with benzocaine paste (Test condom A and Test condom B) will be evaluated against a standard NRL male condom (Control condom) in prolonging time to ejaculation in healthy adult men who feel they ejaculate too quickly during vaginal sex.

ELIGIBILITY:
Main Inclusion Criteria:

1. Subjects and their female partners have provided written informed consent.
2. Subjects and their female partners between the ages of >= 18 years and =< 60 years.
3. Subjects and their female partners must have no health condition in their medical history.
4. Subject must be sexually active having regular intercourse.
5. Subjects in a stable, monogamous, sexual relationship with the same female partner for more than or equal to 3 months.
6. Subject's female partner should already be on an established other highly effective form of non-barrier contraception, unless post-menopausal.
7. Subjects reporting a frequency of 'occasionally' to the Sexual Intercourse Self-Estimation Scale.

Main Exclusion Criteria:

1. Subject with a pregnant or breastfeeding female partner or the female partner desires to become pregnant during the clinical investigation.
2. Subject or his female partner with a current history of alcohol or drug abuse.
3. Subjects and their female partners with a history of or are suffering from anemia, coronary artery disease, impaired cardiac conduction, pulmonary disease, diabetes, and renal or hepatic disease.
4. Subjects and their female partners with a history of, suspected to have, or be at increased risk of methaemoglobinemia / complications related to ester anaesthetics which could trigger methemoglobinemia.
5. Subject and/or his female partner have a physical or psychological condition that would prevent them from following investigation procedures - including but not limited to the following:

   1. urological disease,
   2. ongoing significant psychiatric disorder not controlled by medication
   3. history of surgery or injury to the pelvis, retroperitoneal surgery, radiotherapy, multiple sclerosis, spinal cord injury, chronic inflammation of the prostate or urethra
   4. relevant previous or planned genital surgery
   5. female partner that has been diagnosed with or treated for vaginal complaints (including vaginal dryness)
   6. any broken skin or wounds in the genital area.
6. Subjects on medication that is contraindicated, which may affect erection.
7. Subject and/or his female partner have any medication which may affect the safety of the subject, including but not limited to benzocaine drug interactions such as cholinesterase inhibitors.
8. Subject and/or his female partner is using or intends to continue to use antibiotics of the sulphonamide type.
9. Subject with premature ejaculation, erectile dysfunction, hypo or hyperthyroidism, hypogonadism, hyperprolactinemia, ejaculatory dysfunction, haemorrhagic disorder, hepatitis B or C, human immunodeficiency virus (HIV) infection or having had penile implant surgery.
10. Subject that has been diagnosed or received treatment for PE (premature ejaculation).
11. Subjects with confirmed erectile dysfunction, hypo or hyperthyroidism, hypogonadism, hyperprolactinemia.
12. Confirmed diagnosis of male subjects with other forms of ejaculatory dysfunction.
13. Subjects that have had prior genital, prostatic or lower tract surgery.
14. Subjects with haemorrhagic disorder, hepatitis B or C, HIV infection or having had penile implant surgery, at any time in their past.
15. Either partner needed to use condoms for a specific STI protection.
16. Subjects and their female partners who have any relevant history of allergy including local anaesthetics, parabens, PABA, commercial hair dyes, paraphenylenediamine, lubricants and latex.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
To determine the effectiveness of benzocaine of the Test Condom A compared with the Control NRL Condom at prolonging time to ejaculation | 4 weeks for each assessment period (intervention duration)
  Subjects will be recording the duration (time in minutes:seconds) from vaginal entry to ejaculation for each condom use. The outcome is evaluated by the change from baseline with the Test Condom A compared to the Control NRL Condom, over a 4-week assessment period.

SECONDARY OUTCOMES:
To determine the effectiveness of benzocaine of the Test Condom B compared with the Control NRL Condom at prolonging time to ejaculation | 4 weeks for each assessment period (intervention duration)
  Subjects will be recording the duration (time in minutes:seconds) from vaginal entry to ejaculation for each condom use. The outcome is evaluated by the change from baseline with the Test Condom B compared to the Control NRL Condom, over a 4-week assessment period.
To determine the effectiveness of benzocaine of the Test Condom A and Test Condom B compared with the Control NRL Condom at prolonging time to ejaculation for an increase of 2, 3 and 4 minutes | 4 weeks for each assessment period (intervention duration)
  Subjects will be recording the duration (time in minutes:seconds) from vaginal entry to ejaculation for each condom use. The outcome is evaluated by the proportion of subjects who achieve an increase of 2, 3 and 4 minutes from baseline in each of the Test Condom A and Test Condom B compared to the Control NRL Condom.
To evaluate the sexual pleasure when using the Test Condom A or Test Condom B compared with the Control NRL Condom | 4 weeks for each assessment period (intervention duration)
  The outcome is assessed by the measure of EMSEX (Event-level Male Sexual) pleasure scale questionnaire, a subject perceived questionnaire, at the end of a 4-week assessment period when using Test Condom A or Test Condom B compared with the Control NRL Condom.
  EMSEX pleasure scale is a 11-item scale which assesses sexual pleasure at the event level. For each item, the range spans the entirety of the potential range from 0 (zero) to 100 (one hundred).
To evaluate the subject's improvement at "lasting longer" for both the Test Condom A and Test Condom B compared with the Control NRL Condom | 4 weeks for each assessment period (intervention duration)
  The outcome is assessed by the measure of Patient Global Impression of Change (PGIC), a subject perceived questionnaire, at the end of a 4-week assessment period when using Test Condom A or Test Condom B compared with the Control NRL Condom. The PGIC is a 7-point response scale (Very much better, Better, Little better, No change, Little worse, Worse, Very much worse).
Subject's experience on the use of each type of condoms [Acceptability and In-Use Tolerability] | 4 weeks for each assessment period (intervention duration)
  Acceptability and in-use tolerability as assessed by subject perceived questionnaires
Total clinical failure rate of each type of condoms | 4 weeks for each assessment period (intervention duration)
  Number of clinical failure events (clinical slippage or clinical breakage) reported by subjects.
Overall proportion of subjects with Adverse Events/Adverse Device Effects (AE/ADEs) | 19 weeks
  Overall proportion of subjects with Adverse Events/Adverse Device Effects (AE/ADEs) i.e. the occurrence of one of more AE/ADE per subject

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin Deuble-Bente, Medical Doctor, Principal Investigator — SGS proderm GmbH
Locations (1):
- SGS proderm GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
IPD will be shared as per local regulations.